CLINICAL TRIAL: NCT06826118
Title: A Single-Arm, Multicenter, Prospective, Exploratory Clinical Study of Axicabtagene Ciloleucel Injection in Patients With Relapsed/Refractory Follicular Lymphoma
Brief Title: Axicabtagene Ciloleucel Injection in Patients With Relapsed/Refractory Follicular Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Bing, Xu, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-16
Record Dates: First submitted 2025-02-10; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Lymphoma; Follicular Lymphoma; Refractory Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — axicabtagene ciloleucel

STUDY DESIGN:
Intervention Model Description: Axicabtagene Ciloleucel Injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Axicabtagene Ciloleucel Injection (Experimental): The total blood volume circulated is recommended to be approximately 8-10 liters to obtain about (5-10)×10^9 mononuclear cells. The collected sample will be packaged according to the study product manual and quickly transported to the cell preparation center for the preparation of Axicabtagene Ciloleucel Injection.
  Pre-treatment chemotherapy. Axicabtagene Ciloleucel Injection infusion.
  Interventions: Drug: Axicabtagene Ciloleucel

INTERVENTIONS:
Drug: Axicabtagene Ciloleucel — Pre-treatment chemotherapy: Cyclophosphamide 500 mg/m² and Fludarabine 30 mg/m² will be administered intravenously on Days -5, -4, and -3 (with the day of Axicabtagene Ciloleucel Injection infusion being Day 0).
  Axicabtagene Ciloleucel Injection infusion: A single dose of autologous T cells transduced with chimeric antigen receptor (CAR) in the form of Axicabtagene Ciloleucel Injection will be administered to the subject intravenously. The target dose is 2.0×10^6 anti-CD19 CAR-T cells/kg body weight. The minimum dose that can be used is 1.5×10^6 anti-CD19 CAR-T cells/kg body weight. For subjects with a body weight of ≥100 kg, the maximum total dose is 2.0×10^8 anti-CD19 CAR-T cells
  Other Names: Axicabtagene Ciloleucel Injection

SUMMARY:
A prospective collection of data on the treatment of Chinese patients with relapsed/refractory follicular lymphoma (FL) using Axicabtagene Ciloleucel Injection, and evaluation of the efficacy and safety of Axicabtagene Ciloleucel Injection in this treatment.

DETAILED DESCRIPTION:
This study is a single-arm, multicenter, prospective Phase II clinical trial, planning to enroll 30 Chinese subjects with relapsed/refractory follicular lymphoma (R/R FL) who will receive Axicabtagene Ciloleucel Injection. The study aims to assess the efficacy and safety of Axicabtagene Ciloleucel Injection in treating Chinese patients with R/R FL.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed follicular lymphoma (FL) grade 1, 2, or 3a according to WHO 2016 classification criteria
2. Subjects with relapsed or refractory FL after prior second-line or higher therapy Prior therapy must include: anti-CD20 monoclonal antibody in combination with an alkylating agent (anti-CD20 monoclonal antibody monotherapy is not eligible as a line of therapy for eligibility). Subjects who have had stable disease (no recurrence) for more than 1 year after completion of their last treatment do not meet the enrollment criteria Translated with DeepL.com (free version)
3. At least one measurable lesion according to the Lugano 2014 classification (Cheson 2014). Lesions with prior radiotherapy were considered measurable only if definitive progression was confirmed after completion of radiotherapy.
4. Patients with FL lymphoma secondary to central may be included in the
5. Previous systemic therapy at least 2 weeks or 5 half-lives (whichever is shorter) from the start of leukapheresis, except for immune checkpoint inhibitors/agonists; Systemic immune checkpoint inhibitor/agonist therapy at least 3 half-lives from leukapheresis (e.g., Ipilimumab, Ivolumab, Pembrolizumab, Atezolizumab, OX40 agonist, 4-IBB agonist). Atezolizumab, OX40 agonist, 4-IBB agonist)
6. Toxic reactions from prior anti-lymphoma therapy must stabilize and recover to ≤ grade 1 (except for non-clinically significant toxicities such as alopecia/balding)
7. ≥ 18 years old
8. ECOG physical status score of 0 or 1
9. Absolute neutrophil count (ANC) ≥ 1.0×10^9/L
10. Platelet count ≥ 75×10^9/L
11. Absolute lymphocyte count ≥ 0.1×10^ 9/L
12. Adequate renal, hepatic, pulmonary, and cardiac function, defined as: 1) total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN), except in subjects with Gilbert's syndrome; 2) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN 3) serum creatinine (Cr) ≤ 1.5 x ULN or creatinine clearance (CCr) ≥ 60 mL/min, with creatinine clearance estimated based on the cockcroft-Gault formula; 4) cardiac ejection fraction ≥ 50%, absence of pericardial effusion as determined by echocardiography (ECHO), and absence of clinically significant cardiac arrhythmia; 5) baseline transcutaneous oxygen saturation > 92% under room ventilation; 6) absence of clinically significant chest pain; and ) absence of clinically significant pleural effusion.
13. A negative serum pregnancy test is required for women of childbearing potential (women who have been surgically sterilized or who are at least 2 years postmenopausal are not considered to be of childbearing potential).

Exclusion Criteria:

1. Converted FL
2. Small lymphocytic lymphoma
3. The histologic grading of FL was 3b
4. lymphoplasmacytic lymphoma
5. Subject has had other malignant tumors unless he/she has survived disease-free and has not received antitumor therapy for at least 3 years; except for non-melanoma skin tumors, carcinoma in situ (e.g., cervix, bladder, breast)
6. Autologous Hematopoietic Stem Cell Transplantation Within 6 Weeks Prior to Scheduled Infusion of Achille's Bromide Injection
7. Has performed allogeneic hematopoietic stem cell transplants
8. Previous CD19-targeted therapy
9. Previous chimeric antigen receptor cell therapy or other genetically modified T-cell therapy.
10. History of severe rapid-onset hypersensitivity reactions to aminoglycosides
11. Presence or suspicion of uncontrolled fungal, bacterial, viral or other infections that require intravenous drug therapy
12. Known human immunodeficiency virus (HIV) infection or active acute or chronic hepatitis infection (HBV or HCV). Subjects with a history of hepatitis must undergo standard serologic or genetic testing in accordance with the most recent version of clinical guidelines/institutional protocols to confirm resolution of infection prior to enrollment.
13. Known history of lymphoma involving the entire gastric wall
14. Presence of any indwelling tube or catheter (e.g., percutaneous nephrostomy tube, indwelling urinary catheter, indwelling biliary drain, or pleural/peritoneal/pericardial catheter). Dedicated central venous access catheters such as Port-a-Cath or Hickman catheters are permitted.
15. Patients with primary central nervous system lymphoma (PCNSL)
16. Subjects with lymphomatous infiltration of the atria or ventricles
17. Myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris, congestive heart failure class II or worse according to the New York Heart Association cardiac classification, or other clinically significant cardiac disease within 12 months prior to enrollment
18. Anticipated emergencies requiring urgent treatment due to rapid tumor progression within 6 weeks of leukapheresis (e.g., tumor mass compression, tumor lysis syndrome)
19. End-organ damage due to autoimmune disease (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) within the past 2 years, or systemic use of immunosuppressive or other systemic disease-control medications. Subjects with a history of autoimmune hypothyroidism who are on a stable dose of thyroid replacement hormone therapy and type I diabetes mellitus on a stable insulin regimen are eligible for enrollment in this study.
20. History of symptomatic deep vein thrombosis (DVT) or pulmonary embolism within 6 months prior to enrollment and history of DVT at the end of the upper extremity within 3 months prior to pretreatment chemotherapy
21. Any medical condition that may affect the assessment of safety or efficacy
22. Has had a severe rapid-onset hypersensitivity reaction to any of the drugs to be used in this study
23. Live, attenuated vaccines administered within ≤6 weeks prior to the start of the pretreatment regimen or whose use is expected to be required during the course of the study;
24. Women of childbearing age who are breastfeeding
25. Male or female subjects who are unwilling to use contraception from the date of signed informed consent until 6 months after completion of pretreatment chemotherapy, or 6 months after completion of an infusion of Aquilensa
26. Male or female subjects who are unwilling to use contraception from the date of signed informed consent until 6 months after completion of pretreatment chemotherapy, or 6 months after completion of an infusion of Aquilensa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Best Objective Response Rate (bORR) at 6 months | Up to 36 months
  This is defined as the proportion of subjects in the modified Intent-To-Treat (mITT) analysis set who achieve a best response of Complete Remission (CR) or Partial Remission (PR) following infusion of Axicabtagene Ciloleucel Injection, as determined by the treating physician, and who have the opportunity to complete the 6-month assessment. Before the data cutoff date, all subjects who do not meet the criteria for objective response will be considered as having no objective response (e.g., those without valid assessments or who did not undergo efficacy evaluation).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 36 months
  Defined as the time interval from the date of Axicabtagene Ciloleucel Injection infusion to the date of disease progression or death due to any cause (whichever occurs first) in the modified Intent-To-Treat (mITT) analysis set.
Complete Response (CR) Rate | Up to 36 months
  Defined as the proportion of subjects in the modified Intent-To-Treat (mITT) analysis set who achieve a best response of Complete Response (CR) as determined by the treating physician.
Partial Response (PR) Rate | Up to 36 months
  Defined as the proportion of subjects in the modified Intent-To-Treat (mITT) analysis set who achieve a best response of Partial Response (PR) as determined by the treating physician.
Duration of Response (DOR) | Up to 36 months
  Defined as the time interval from the first documented complete or partial response to disease progression or death due to any cause (whichever occurs first) among subjects who achieve an objective response in the modified Intent-To-Treat (mITT) analysis set.
Overall Survival (OS) | Up to 36 months
  Defined as the time interval from the infusion of Axicabtagene Ciloleucel Injection to death due to any cause in the modified Intent-To-Treat (mITT) analysis set. All subjects, regardless of whether they receive any additional anti-tumor treatment after infusion, will be followed up for survival information. The causes of death will also be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- Bing Xu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No